CLINICAL TRIAL: NCT00725894
Title: A Prospective Multi-Center Clinical Outcomes Study To Assess The Safety and Effectiveness Of The Pediatric Locking Nail For Treatment Of Femoral Fractures In Children
Brief Title: Pediatric Locking Nail for the Treatment of Femoral Fractures in Children
Acronym: PLN
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-010
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The Pediatric Locking Nail was designed to provide stable sub-rigid fixation of femoral fractures in children
  Interventions: Device: Pediatric Locking Nail

INTERVENTIONS:
Device: Pediatric Locking Nail — The nail is pre contoured with a nine-degree anterior bow and is universal for right and left femoral.

SUMMARY:
The purpose of this multi-center prospective clinical outcomes study is to determine validity and safety of the pediatric locking nail for femoral fracture management in children with open physes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, representative willing to sign informed consent.
2. Ability and willingness of the subject to follow postoperative care instructions until healing is complete
3. Subject age must be between 8-16 inclusive.
4. Subjects with a minimal canal diameter of 9mm or greater

And any of the following fracture types

1. Non-comminuted and comminuted mid-shaft fractures
2. Distal third fractures 4 cm above the distal physis
3. Fractures that are open or closed
4. Subtrochanteric fractures

Exclusion Criteria:

1. A subject has a bone or soft tissue infection.
2. Subject has a systemic infection.
3. Subject has a distal (supracondylar) fracture.
4. Subject with pathological bone (osteogenesis imperfecta and other conditions resulting in abnormal bone quality).
5. Subjects with mental or neurological condition who are unwilling or incapable of following postoperative care instructions.
6. Subject with conditions including blood supply limitation, and insufficient quantity or quality of bone.
7. Foreign body sensitivity, where material sensitivity is suspected, testing is to be completed prior to implantation of device if at all practical or the subject should be excluded.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric femoral fractures in patients 8-16 years of age where a nail is preferred
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
limb alignment | 48 months

SECONDARY OUTCOMES:
length of healing, weight-bearing time (time to full weight bearing), and length of hospital stay and absence of complications | 48 Months

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, PhD, Study Director — Zimmer Biomet
Locations (3):
- United States (3):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arnold Palmer Hospital for Children/OH Pediatric Orthopedics Clinic, Orlando, Florida
  - Orthopedic Clinical Research, Charlotte, North Carolina